CLINICAL TRIAL: NCT06255574
Title: Correlation Between Cervical Spine Sagittal Alignment and Functional Disability in Preparatory School Students With Mechanical Cervical Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Manal Helmy Koura, Lecturer, Benha University
Other Study IDs: PT.BU.EC.4
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Children, Only
Keywords: cervical spine; sagittal alignment; functional disability; preparatory school children; mechanical cervical pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neck pain is a major public health concern that has been extensively studied in adults but not in children and adolescents. Mechanical neck pain became prevalent among children and adolescents, and has its impacts on functional ability.

This study is aiming to investigate the correlation between Cervical spine sagittal alignment parameter (cranio-cervical angle) and functional disability in preparatory school students with mechanical cervical pain.

DETAILED DESCRIPTION:
* Correlational study between cranio-cervical angles and functional disability in students with mechanical cervical pain.
* Inclusion Criteria Age between 12 and 15 years, either sex, and cervical symptoms lasting longer than three months.
* exclusion criteria Spinal pathologies or surgery, or any other deformities or visual or auditory issues, as well as ongoing physical or medical treatment for cervical pain

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 15 years, either sex, and cervical symptoms lasting longer than three months.

Exclusion Criteria:

* Spinal pathologies or surgery, or any other deformities or visual or auditory issues, as well as ongoing physical or medical treatment for cervical pain

Ages: 12 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Preparatory school age students
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
● cervico cranial angle by X-ray device | one hour
  ● X-ray device: (Toshiba Rotande unite model DRX3724 HD/2009 will be used.
Functional neck status | one hour
  Functional status will be evaluated by Neck Disability index (NDI).

IPD SHARING:
Plan to Share IPD: No